CLINICAL TRIAL: NCT01209598
Title: A Phase II Study Of PD0332991 (Palbociclib) in Patients With Advanced or Metastatic Liposarcoma
Brief Title: PD0332991 (Palbociclib) in Patients With Advanced or Metastatic Liposarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-094
Record Dates: First submitted 2010-09-24; First posted 2010-09-27 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-02

CONDITIONS: Sarcoma; Liposarcoma
Keywords: soft tissue; Palbociclib (PD0332991); 10-094
MeSH Terms: conditions — Sarcoma; Liposarcoma | interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Palbociclib 200mg (Experimental): This is a phase II study of Palbociclib in patients with advanced / metastatic liposarcoma. A one-stage design is used to determine whether patients treated with Palbociclib achieved a PFS rate of ≥ 40% at 12 weeks.
  Interventions: Drug: Palbociclib 200mg
- Palbociclib 125mg (Experimental): This is a phase II study of Palbociclib in patients with advanced / metastatic liposarcoma. A one-stage design is used to determine whether patients treated with Palbociclib achieved a PFS rate of ≥ 40% at 12 weeks.
  Interventions: Drug: Palbociclib 125mg

INTERVENTIONS:
Drug: Palbociclib 200mg — Schedule 2/1: Palbociclib 200mg given once daily by mouth for 14 consecutive days, followed by 7 days of rest. A cycle will be defined as 21 days.
  Arms: Palbociclib 200mg
Drug: Palbociclib 125mg — Schedule 3/1: Palbociclib 125mg given once daily by mouth for 21 consecutive days, followed by 7 days of rest. A cycle will be defined as 28 days. Following the positive results of the study, a new Expansion Cohort has been added to permit enrollment of up to 20 additional patients.
  Expansion Cohort: Dosed as per Schedule 3/1. Capsules should be taken with food.
  Arms: Palbociclib 125mg

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, Palbociclib (Ibrance) (formerly known as PD0332991) has on the patient and on the liposarcoma.

Palbociclib is an investigational drug. An investigational drug is a medication that has not been approved for marketing by the Food and Drug Administration (FDA). Palbociclib blocks a protein called CDK4 which is part of a pathway in liposarcoma cells that is over-active. The investigators hope that blocking CDK4 will shut down this pathway in the liposarcoma cells and stop tumors from growing. Palbociclib is an oral medication.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of liposarcoma confirmed at MSKCC. Because myxoid / round cell liposarcoma does not have significant CDK4 amplification, patients with this subtype are not eligible.
* Metastatic and/or locally advanced or locally recurrent disease that is not surgically resectable, with evidence of disease progression, either clinically or radiographically, as determined by the investigator
* All patients must have measurable disease as defined by RECIST 1.1. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded). Each lesion must be >10 mm when measured by CT, MRI or caliper measurement by clinical exam; or >20 mm when measured by chest x-ray. Lymph nodes must be > 15 mm in short axis when measured by CT or MRI.
* A minimum of 1 prior systemic regimen for recurrent/metastatic disease. Note: This requirement does not apply to patients enrolled in the Expansion Cohort. The last dose of systemic therapy (include targeted therapies) must have been given at least 2 weeks prior to initiation of therapy. Patients receiving BCNU or mitomycin C must have received their last dose of such therapy at least 6 weeks prior to initiation of therapy.
* Patients with brain metastasis that have been treated with definitive surgery or radiation and have been clinically stable for 3 months are eligible.
* Age > or = 18 years.
* ECOG performance status 0 or 1.
* Adequate organ and marrow function as defined below (ULN indicates institutional upper limit of normal):

Absolute neutrophil count ≥ 1.5x109/L Hemoglobin ≥ 9.0 g/dL WBC ≥ 3.0x109/L Platelets ≥ 100x109/L Total bilirubin ≤ 1.5 x ULN except for patients with known Gilbert syndrome AST(SGOT)/ALT(SGPT) ≤ 3 x institutional ULN Serum creatinine ≤ 1.5 x ULN or Creatinine Clearance > 50 mL/min (calculated by Cockcroft-Gault method)QTc interval ≤ 470 msec

* Patients must not have current evidence of another malignancy that requires treatment.
* The effects of Palbociclib on the developing human fetus at the recommended therapeutic dose are unknown. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence). Women must not breast feed while on study.
* Ability to understand and the willingness to sign a written informed consent document.
* Ability to swallow intact Palbociclib capsules.
* Patients" tumors must express Rb, as assessed using an historical biopsy sample if available or a newly obtained tumor sample. Samples must demonstrate ≥1+ staining for Rb. Patients' tumors must also have evidence of CDK4 amplification by FISH. Note: This does not apply to patients enrolled in the Expansion Cohort.

Exclusion Criteria:

* Patients who have not recovered from adverse events of prior therapy to ≤ NCI CTCAEv4.0 Grade 1.
* Patients receiving any other investigational agents.
* Patients who have received prior treatment with a selective CDK4 inhibitor
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Palbociclib.
* Uncontrolled intercurrent illness including, but not limited to, known ongoing or active infection, including HIV, active hepatitis B or C, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia (specifically, atrial fibrillation or ventricular dysrhythmias except ventricular premature contractions), or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women and women who are breast-feeding.
* Patients with a history of long-QT syndrome or documented family history of long-QT syndrome. Patients who must remain on drugs that prolong the QT interval.
* Palbociclib is a substrate of CYP3A. Caution should be exercised when dosing Palbociclib concurrently with CYP3A inducers or inhibitors. Furthermore, patients who are taking concurrent medications that are strong inducers/inhibitors or substrates of CYP3A4 should be switched to alternative medications to minimize any potential risk. A list of CYP3A4 substrates, inducers and/or inhibitors is provided in Appendix B. The following medications with strong potential for interaction are not allowed: indinavir nelfinavir ritonavir clarithromycin itraconazole ketoconazole nefazodone saquinavir telithromycin carbamazepine phenobarbital phenytoin pioglitazone rifabutin rifampin St. John's wort Troglitazone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-09-23 (Actual); Primary Completion 2016-10-25 (Actual); Study Completion 2016-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Dickson, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] McAndrew NP, Dickson MA, Clark AS, Troxel AB, O'Hara MH, Colameco C, Gallager M, Gramlich K, Zafman K, Vaughn D, Schwartz GK, O'Dwyer PJ, DeMichele A. Early treatment-related neutropenia predicts response to palbociclib. Br J Cancer. 2020 Sep;123(6):912-918. doi: 10.1038/s41416-020-0967-7. Epub 2020 Jul 9. PMID 32641862
- [Derived] Dickson MA, Schwartz GK, Keohan ML, D'Angelo SP, Gounder MM, Chi P, Antonescu CR, Landa J, Qin LX, Crago AM, Singer S, Koff A, Tap WD. Progression-Free Survival Among Patients With Well-Differentiated or Dedifferentiated Liposarcoma Treated With CDK4 Inhibitor Palbociclib: A Phase 2 Clinical Trial. JAMA Oncol. 2016 Jul 1;2(7):937-40. doi: 10.1001/jamaoncol.2016.0264. PMID 27124835
- [Derived] Dickson MA, Tap WD, Keohan ML, D'Angelo SP, Gounder MM, Antonescu CR, Landa J, Qin LX, Rathbone DD, Condy MM, Ustoyev Y, Crago AM, Singer S, Schwartz GK. Phase II trial of the CDK4 inhibitor PD0332991 in patients with advanced CDK4-amplified well-differentiated or dedifferentiated liposarcoma. J Clin Oncol. 2013 Jun 1;31(16):2024-8. doi: 10.1200/JCO.2012.46.5476. Epub 2013 Apr 8. PMID 23569312
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual 09/23/2010 Protocol Closed to Accrual 05/27/2014 Primary Completion Date 10/25/2016 Recruitment Location is the medical clinic
Groups:
- Palbociclib 125mg: This is a phase II study of Palbociclib in patients with advanced / metastatic liposarcoma. A one-stage design is used to determine whether patients treated with Palbociclib achieved a PFS rate of ≥ 40% at 12 weeks.
  Palbociclib 125mg: Schedule 3/1: Palbociclib 125mg given once daily by mouth for 21 consecutive days, followed by 7 days of rest. A cycle will be defined as 28 days. Following the positive results of the study, a new Expansion Cohort has been added to permit enrollment of up to 20 additional patients.
Period: Overall Study
Arm/Group | Palbociclib 200mg | Palbociclib 125mg
Started | 30 | 60
Completed | 29 | 60
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Palbociclib 200mg | Palbociclib 125mg | Total
Number analyzed (Participants) | 30 | 60 | 90
Age, Continuous [Median (Full Range); unit: years] | 65 [37 to 83] | 61.5 [35 to 87] | 62 [35 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 31 | 47
  Male | 14 | 29 | 43
Region of Enrollment [Number; unit: participants]
  United States | 30 | 60 | 90

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival at 12 Weeks
Description: PFS, defined as RECIST 1.1 (CR + PR + SD) when treated with Palbociclib
Time Frame: 12 weeks
Measure: Median (95% Confidence Interval); unit: percentage of particpants
Arm/Group | Palbociclib 200mg | Palbociclib 125mg
Number analyzed (Participants) | 30 | 60
percentage of particpants | 66 [51 to 100] | 57.2 [42.4 to 68.8]

2. Secondary Outcome: Best Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Palbociclib 125mg: This is a phase II study of Palbociclib in patients with advanced / metastatic liposarcoma. A one-stage design is used to determine whether patients treated with Palbociclib achieved a PFS rate of ≥ 40% at 12 weeks.
  Palbociclib 125mg: Schedule 3/1: Palbociclib 125mg given once daily by mouth for 21 consecutive days, followed by 7 days of rest. A cycle will be defined as 28 days. Following the positive results of the study, a new Expansion Cohort has been added to permit enrollment of up to 20 additional patients.
  Expansion Cohort: Dosed as per Schedule 3/1. Capsules should be taken with food.
Arm/Group | Palbociclib 200mg | Palbociclib 125mg
Number analyzed (Participants) | 30 | 60
Participants
  Partial Response | 1 | 0
  Complete Response | 0 | 1
  Stable Disease | 5 | 8
  Progression of Disease | 23 | 50
  Non-Evaluable | 1 | 1

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Palbociclib 200mg | Palbociclib 125mg
Serious Adverse Events (participants affected / at risk) | 24/30 | 55/60
Other Adverse Events (participants affected / at risk) | 30/30 | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palbociclib 200mg (N=30) | Palbociclib 125mg (N=60)
Constipation (Gastrointestinal disorders) | 1 | 0
Death NOS (General disorders) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0
Fatigue (General disorders) | 2 | 0
Anemia (Blood and lymphatic system disorders) | 5 | 13
Lymphocyte count decreased (Investigations) | 9 | 19
Platelet count decreased (Investigations) | 9 | 4
White blood cell decreased (Investigations) | 14 | 15
Neutrophil count decreased (Investigations) | 15 | 22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Palbociclib 200mg (N=30) | Palbociclib 125mg (N=60)
Anorexia (Metabolism and nutrition disorders) | 2 | 0
Dizziness (Nervous system disorders) | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Edema limbs (General disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Skin & subcutaneous tissue disorders Other, spec (Skin and subcutaneous tissue disorders) | 2 | 0
Fever (General disorders) | 3 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 0
Musculoskeletal & conn tissue disorder Other, spec (Musculoskeletal and connective tissue disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 4 | 3
Constipation (Gastrointestinal disorders) | 5 | 0
Diarrhea (Gastrointestinal disorders) | 6 | 4
Nausea (Gastrointestinal disorders) | 8 | 10
Lymphocyte count decreased (Investigations) | 9 | 13
Mucositis oral (Gastrointestinal disorders) | 9 | 7
Fatigue (General disorders) | 14 | 15
Anemia (Blood and lymphatic system disorders) | 24 | 55
Platelet count decreased (Investigations) | 25 | 35
Neutrophil count decreased (Investigations) | 26 | 45
White blood cell decreased (Investigations) | 28 | 57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-13): https://cdn.clinicaltrials.gov/large-docs/98/NCT01209598/Prot_SAP_000.pdf